CLINICAL TRIAL: NCT04405908
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, First-in-human Study to Evaluate the Safety and Immunogenicity of SCB 2019, a Recombinant SARS-CoV-2 Trimeric S Protein Subunit Vaccine for COVID-19 in Healthy Volunteers.
Brief Title: SCB-2019 as COVID-19 Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clover Biopharmaceuticals AUS Pty (Industry)
Responsible Party: Sponsor
Organization: Clover Biopharmaceuticals, Ltd (Industry)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: CLO-SCB-2019-001
Record Dates: First submitted 2020-05-25; First posted 2020-05-28 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — SCB-2019 COVID-19 vaccine; AS03 adjuvant; Aluminum Hydroxide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (27):
- Adult Group 1 (Placebo Comparator): Adult healthy subjects (18 to 54 years of age, inclusive) receive SCB-2019 3 µg.
  Interventions: Biological: SCB-2019
- Adult Group 2 (Placebo Comparator): Adult healthy subjects (18 to 54 years of age, inclusive) receive SCB-2019 3 µg with AS03 adjuvant.
  Interventions: Biological: SCB-2019 with AS03 adjuvant
- Adult Group 3 (Placebo Comparator): Adult healthy subjects (18 to 54 years of age, inclusive) receive SCB-2019 3 µg with CpG 1018 plus Alum adjuvant.
  Interventions: Biological: SCB-2019 with CpG 1018 adjuvant plus Alum adjuvant
- Adult Group 4 (Placebo Comparator): Adult healthy subjects (18 to 54 years of age, inclusive) receive SCB-2019 9 µg .
  Interventions: Biological: SCB-2019
- Adult Group 5 (Placebo Comparator): Adult healthy subjects (18 to 54 years of age, inclusive) receive SCB-2019 9 µg with AS03 adjuvant.
  Interventions: Biological: SCB-2019 with AS03 adjuvant
- Adult Group 6 (Placebo Comparator): Adult healthy subjects (18 to 54 years of age, inclusive) receive SCB-2019 9 µg with CpG 1018 plus Alum adjuvant.
  Interventions: Biological: SCB-2019 with CpG 1018 adjuvant plus Alum adjuvant
- Adult Group 7 (Placebo Comparator): Adult healthy subjects (18 to 54 years of age, inclusive) receive SCB-2019 30 µg .
  Interventions: Biological: SCB-2019
- Adult Group 8 (Placebo Comparator): Adult healthy subjects (18 to 54 years of age, inclusive) receive SCB-2019 30 µg with AS03 adjuvant.
  Interventions: Biological: SCB-2019 with AS03 adjuvant
- Adult Group 9 (Placebo Comparator): Adult healthy subjects (18 to 54 years of age, inclusive) receive SCB-2019 30 µg with CpG 1018 plus Alum adjuvant.
  Interventions: Biological: SCB-2019 with CpG 1018 adjuvant plus Alum adjuvant
- Elderly Group 10 (Placebo Comparator): Elderly healthy subjects (55 to 75 years of age, inclusive) receive SCB-2019 3 µg with AS03 adjuvant.
  Interventions: Biological: SCB-2019 with AS03 adjuvant
- Elderly Group 11 (Placebo Comparator): Elderly healthy subjects (55 to 75 years of age, inclusive) receive SCB-2019 3 µg with CpG 1018 plus Alum adjuvant.
  Interventions: Biological: SCB-2019 with CpG 1018 adjuvant plus Alum adjuvant
- Elderly Group 12 (Placebo Comparator): Elderly healthy subjects (55 to 75 years of age, inclusive) receive SCB-2019 9 µg with AS03 adjuvant.
  Interventions: Biological: SCB-2019 with AS03 adjuvant
- Elderly Group 13 (Placebo Comparator): Elderly healthy subjects (55 to 75 years of age, inclusive) receive SCB-2019 9 µg with CpG 1018 plus Alum adjuvant.
  Interventions: Biological: SCB-2019 with CpG 1018 adjuvant plus Alum adjuvant
- Elderly Group 14 (Placebo Comparator): Elderly healthy subjects (55 to 75 years of age, inclusive) receive SCB-2019 30 µg with AS03 adjuvant.
  Interventions: Biological: SCB-2019 with AS03 adjuvant
- Elderly Group 15 (Placebo Comparator): Elderly healthy subjects (55 to 75 years of age, inclusive) receive SCB-2019 30 µg with CpG 1018 plus Alum adjuvant.
  Interventions: Biological: SCB-2019 with CpG 1018 adjuvant plus Alum adjuvant
- SARS-CoV-2 Seropositive Group 16 (Placebo Comparator): SARS-CoV-2 Seropositive subjects receive SCB-2019 9 µg.
  Interventions: Biological: SCB-2019
- SARS-CoV-2 Seropositive Group 17 (Placebo Comparator): SARS-CoV-2 Seropositive subjects receive SCB-2019 9 µg with AS03 adjuvant.
  Interventions: Biological: SCB-2019 with AS03 adjuvant
- SARS-CoV-2 Seropositive Group 18 (Placebo Comparator): SARS-CoV-2 Seropositive subjects receive SCB-2019 30 µg with CpG 1018 plus Alum adjuvant.
  Interventions: Biological: SCB-2019 with CpG 1018 adjuvant plus Alum adjuvant
- Adjuvant Dose Modification: Adult Group 19 (Placebo Comparator): Adult healthy subjects (18 to 54 years of age, inclusive) receive SCB-2019 9 µg with AS03 adjuvant.
  Interventions: Biological: SCB-2019 with AS03 adjuvant
- Adjuvant Dose Modification: Adult Group 20 (Placebo Comparator): Adult healthy subjects (18 to 54 years of age, inclusive) receive SCB-2019 30 µg with CpG 1018 plus Alum adjuvant.
  Interventions: Biological: SCB-2019 with CpG 1018 adjuvant plus Alum adjuvant
- Adjuvant Dose Modification: Elderly Group 21 (Placebo Comparator): Elderly healthy subjects (55 to 75 years of age, inclusive) receive SCB-2019 9 µg with AS03 adjuvant.
  Interventions: Biological: SCB-2019 with AS03 adjuvant
- Adjuvant Dose Modification: Elderly Group 22 (Placebo Comparator): Elderly healthy subjects (55 to 75 years of age, inclusive) receive SCB-2019 30 µg with CpG 1018 plus Alum adjuvant.
  Interventions: Biological: SCB-2019 with CpG 1018 adjuvant plus Alum adjuvant
- Alum Only Adjuvant Group 23 (Placebo Comparator): Subjects receive SCB-2019 9 µg with Alum adjuvant only.
  Interventions: Biological: SCB-2019 with Alum adjuvant
- Dose Expansion Phase: Adult Group 24 (Placebo Comparator): Adult healthy subjects (18 to 54 years of age, inclusive) receive SCB-2019 9 µg with AS03 adjuvant.
  Interventions: Biological: SCB-2019 with AS03 adjuvant
- Dose Expansion Phase: Adult Group 25 (Placebo Comparator): Adult healthy subjects (18 to 54 years of age, inclusive) receive SCB-2019 30 µg with CpG 1018 plus Alum adjuvant.
  Interventions: Biological: SCB-2019 with CpG 1018 adjuvant plus Alum adjuvant
- Dose Expansion Phase: Elderly Group 26 (Placebo Comparator): Elderly healthy subjects (55 to 75 years of age, inclusive) receive SCB-2019 9 µg with AS03 adjuvant.
  Interventions: Biological: SCB-2019 with AS03 adjuvant
- Dose Expansion Phase: Elderly Group 27 (Placebo Comparator): Elderly healthy subjects (55 to 75 years of age, inclusive) receive SCB-2019 30 µg with CpG 1018 plus Alum adjuvant.
  Interventions: Biological: SCB-2019 with CpG 1018 adjuvant plus Alum adjuvant

INTERVENTIONS:
Biological: SCB-2019 — SCB-2019 intramuscular vaccinations at 3 µg up to 30 µg twice (on Day 1 and Day 22).
  Arms: Adult Group 1; Adult Group 4; Adult Group 7; SARS-CoV-2 Seropositive Group 16
Biological: SCB-2019 with AS03 adjuvant — SCB-2019 intramuscular vaccinations at 3 µg up to 30 µg twice (on Day 1 and Day 22), and administered with AS03 adjuvant.
  Arms: Adjuvant Dose Modification: Adult Group 19; Adjuvant Dose Modification: Elderly Group 21; Adult Group 2; Adult Group 5; Adult Group 8; Dose Expansion Phase: Adult Group 24; Dose Expansion Phase: Elderly Group 26; Elderly Group 10; Elderly Group 12; Elderly Group 14; SARS-CoV-2 Seropositive Group 17
Biological: SCB-2019 with CpG 1018 adjuvant plus Alum adjuvant — SCB-2019 intramuscular vaccinations at 3 µg up to 30 µg twice (on Day 1 and Day 22), and administered with CpG 1018 plus Alum adjuvant.
  Arms: Adjuvant Dose Modification: Adult Group 20; Adjuvant Dose Modification: Elderly Group 22; Adult Group 3; Adult Group 6; Adult Group 9; Dose Expansion Phase: Adult Group 25; Dose Expansion Phase: Elderly Group 27; Elderly Group 11; Elderly Group 13; Elderly Group 15; SARS-CoV-2 Seropositive Group 18
Biological: SCB-2019 with Alum adjuvant — SCB-2019 intramuscular vaccinations at 9 µg twice (on Day 1 and Day 22), and administered with Alum adjuvant.
  Arms: Alum Only Adjuvant Group 23

SUMMARY:
This is a randomized, double blind, placebo controlled, first-in-human (FIH) study to assess safety, reactogenicity, and immunogenicity of SCB-2019 at multiple dose levels, administered as 2 injections IM in healthy subjects. Each study vaccine dose level will be evaluated with and without adjuvant.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or females, ≥18 years of age at Screening:

   1. For the adult group: 18 to 54 years, inclusive, and
   2. For the elderly group: 55 to 75 years, inclusive.
2. Individuals who are willing and able to give an informed consent, prior to Screening.
3. Individuals who are able to comply with study requirements.
4. Female subjects are eligible to participate in the study if not pregnant, not breastfeeding, and at least 1 of the following criteria apply:

   1. Women of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test prior to each vaccination. They must be using a highly effective licensed method of birth control for 30 days prior to the first dose of the study vaccine/placebo and must agree to continue such precautions during the study until 60 days after the second dose of the study vaccine/placebo.
   2. Women not of childbearing potential, defined as surgically sterile (documented hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or postmenopausal (no menses for 12 months and follicle-stimulating hormone [FSH] in the postmenopausal range).
   3. Male subjects must agree to employ acceptable contraception from the day of first dose of the study vaccine/placebo until 90 days after the second dose of the study vaccine/placebo and also refrain from donating sperm during this period.
5. General good health based on medical history, physical examination, cardiac health evaluation, and clinical laboratory evaluations. Participants in the elderly population who have medically stable, well-controlled co-morbidities may be enrolled at the discretion of the Investigator.

   All clinical laboratory values should be within normal reference ranges unless confirmed by Investigator or delegate as not clinically significant. One repeat evaluation of electrocardiogram (ECG), and clinical laboratory tests will be permitted, at the discretion of the Investigator.
6. Individuals agree to avoid strenuous exercise from Screening to Day 50.

   For the SARS-CoV-2 seropositive treatment group only (Treatment Groups 16 to 18):
7. Serological or ELISA confirmation of SARS-CoV-2;
8. No history of severe SARS-CoV-2 symptoms;
9. No SARS-CoV-2 symptoms at the time of the screening .

Exclusion Criteria:

1. Individuals with any positive test for SARS-CoV-2 infection, including but not limited to RT-PCR, at Screening (excluding the SARS-CoV-2 seropositive treatment group [Treatment Groups 16 to 18]).
2. Individuals with positive serology test results for SARS-CoV-2 at Screening (excluding the SARS-CoV-2 seropositive treatment group [Treatment Groups 16 to 18]).
3. Individuals with behavioral or cognitive impairment in the opinion of the Investigator.
4. Individuals with any progressive or severe neurologic disorder, seizure disorder, or history of Guillian-Barré syndrome.
5. Individuals who are not able to comprehend and to follow all required study procedures for the whole period of the study.
6. Individuals with known or suspected impairment of the immune system, such as:

   1. Use of systemic (oral or parenteral) corticosteroids for ≥14 consecutive days within 60 days prior to Day 1. Use of inhaled, intranasal, or topical corticosteroids is allowed.Note: Systemic (oral or parenteral) corticosteroids are also prohibited for 3 weeks after the second dose of the study vaccine/placebo.
   2. Receipt of cancer chemotherapy within 5 years prior to Day 1.
   3. Receipt of immunostimulants or immunosuppressants within 60 days prior to Day 1.
   4. Known HIV or acquired immune deficiency syndrome (AIDS).
   5. Subjects with active or prior documented autoimmune disorder (such as potential immune-mediated diseases [pIMDs]).
   6. Receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivatives within 3 months prior to Day 1 or planned during the full length of the study.
7. Positive serology test results for hepatitis C virus antibody, HIV antibody, and/or hepatitis B virus surface antigen at Screening.
8. Individuals who are pregnant or breastfeeding.
9. Individuals who are allergic to any of the study vaccine/placebo components as outlined in the current SCB 2019 IB.
10. Individuals who have had a malignancy (excluding nonmelanotic skin cancer) or lymphoproliferative disorder within the past 5 years from the date of first administration of the study vaccine/placebo (Day 1).
11. Individuals who have received any other investigational product within 30 days prior to Day 1 or intent to participate in another clinical study at any time during the conduct of this study.
12. Individuals with a body temperature ≥38.0 °C (≥100.4 °F) or any acute illness within 3 days of intended study vaccination.
13. Individuals who have a previous confirmed or suspected illness caused by coronaviruses, SARS-CoV-1, SARS-CoV-2, and Middle East Respiratory Syndrome (MERS)-CoV (excluding the SARS-CoV-2 seropositive treatment group [Treatment Groups 16 to 18]).
14. Individuals who have received any prior vaccine against a coronavirus, including but not limited to SARS-CoV, SARS-CoV-2, MERS-CoV.
15. Individuals who have received any other licensed vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in this study or who are planning to receive any vaccine within 28 days (before or after) the study vaccine/placebos, with the exception of the seasonal influenza vaccine.
16. Presence of uncontrolled chronic pulmonary, cardiovascular, renal, hepatic, neurologic, hematologic or metabolic (including diabetes mellitus) disorders, which would include the potential subject in a high-risk category for SARS CoV 2 infection and/or its complications.
17. Individuals with known bleeding diathesis.
18. Individuals with a body mass index <18.5 kg/m2 or >35.0 kg/m2.
19. Individuals with a history of drug or alcohol abuse within the past 2 years.
20. Individuals with a history of anaphylaxis or angioedema including but not limited to history of anaphylaxis after any vaccine.
21. Individuals with any condition that, in the opinion of the Investigator, would interfere with the primary study objectives or pose additional subject risk.
22. Individuals who are research staff involved with the clinical study or family/household members of research staff.
23. Individuals must not have donated blood for 2 months prior to Day 1 and must agree to not donate blood for 6 months post Day 1 (receipt of first dose of study vaccine).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
Incidence of solicited adverse events (AEs) after vaccination | 7 days after the first or second vaccination.
  To evaluate the safety and reactogenicity profile of adjuvanted and unadjuvanted SCB-2019 in adult and elderly , when administered as 2 intramuscular doses.
Incidence of unsolicited AEs after vaccination | Day 1 to Day 50
  To evaluate the safety and reactogenicity profile of adjuvanted and unadjuvanted SCB-2019 in adult and elderly , when administered as 2 intramuscular doses.
Mean change from Baseline in safety laboratory measures (include hematology, coagulation panel, and serum chemistry) | Day 1 to Day 50
  To evaluate the safety and reactogenicity profile of adjuvanted and unadjuvanted SCB-2019 in adult and elderly , when administered as 2 intramuscular doses.
Incidence of serious AEs (SAEs) and adverse events of special interest (AESIs) | Day 1 to Day 184
  To evaluate the safety and reactogenicity profile of adjuvanted and unadjuvanted SCB-2019 in adult and elderly , when administered as 2 intramuscular doses.
As assessed by serum anti-SCB-2019 IgG antibody titers | Day 1 to Day 184
  Geometric mean titer (GMT). Geometric mean ratio (GMR). Seroconversion rate (SCR).

SECONDARY OUTCOMES:
Immunogenicity( serum anti SARS-CoV-2 neutralizing antibody titers (ACE2 receptor-based) ) | Day 1 to Day 184
  Geometric mean titer (GMT). Geometric mean ratio (GMR). Seroconversion rate (SCR).
Immunogenicity(serum anti SARS-CoV-2 neutralizing antibody titers (cell based) ) | Day 1 to Day 184
  Geometric mean titer (GMT). Geometric mean ratio (GMR). Seroconversion rate (SCR).
Immunogenicity(serum anti SARS-CoV-2 whole virus antibody titers) | Day 1 to Day 184
  Geometric mean titer (GMT). Geometric mean ratio (GMR). Seroconversion rate (SCR).
Antibody kinetics of each SCB 2019 vaccine formulation after first and second doses | Day 1 to Day 184
  Geometric mean titer (GMT). Geometric mean ratio (GMR). Seroconversion rate (SCR).

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research Ltd, Nedlands, Western Australia, Australia

REFERENCES:
- [Derived] Richmond P, Hatchuel L, Dong M, Ma B, Hu B, Smolenov I, Li P, Liang P, Han HH, Liang J, Clemens R. Safety and immunogenicity of S-Trimer (SCB-2019), a protein subunit vaccine candidate for COVID-19 in healthy adults: a phase 1, randomised, double-blind, placebo-controlled trial. Lancet. 2021 Feb 20;397(10275):682-694. doi: 10.1016/S0140-6736(21)00241-5. Epub 2021 Jan 29. PMID 33524311